CLINICAL TRIAL: NCT05562505
Title: A Randomised Controlled Trial of Venovenous ECMO to De-Sedate, Extubate and Mobilise in Hypoxic Respiratory Failure
Brief Title: Trial of Venovenous ECMO to De-Sedate, Extubate and Mobilise in Hypoxic Respiratory Failure
Acronym: REDEEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANZIC-RC/AB002 V2.0
Record Dates: First submitted 2022-09-11; First posted 2022-09-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Ventilation Complication; Hypoxemia; Acute Respiratory Distress Syndrome Due to COVID-19; COVID-19 Respiratory Infection; Pneumonia; Extracorporeal Membrane Oxygenation
Keywords: Intensive Care Unit; ECMO; Extracorporeal Membrane Oxygenation; Mechanical Ventilation; Early ECMO
MeSH Terms: conditions — Hypoxia; Pneumonia | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venovenous ECMO (Active Comparator): Patients allocated to the ECMO strategy be initiated on V-V ECMO and on anticoagulation (blood thinning medication to prevent clot formation) within 24 hours of being allocated into the intervention group. Anticoagulant medication to prevent clot formation will be initiated as per current local practice for each site. Sites are encouraged to use best practice ECMO management that includes de-sedation, extubation, commencement of physiotherapy and rehabilitation,
  Interventions: Other: Venovenous ECMO
- Standard care (No Intervention): Patients allocated to the standard care arm will receive routine intensive care for hypoxic respiratory failure, including mechanical ventilation as per local practices, weaning of sedation and assessment for extubation. Patients who continue to deteriorate will be eligible for initiation of V-V ECMO if they meet the ECMO to rescue lung injury in severe ARDS (EOLIA) criteria: Partial pressures of arterial oxygen (PaO2):Fraction of inspired oxygen (FiO2)<50 for 3 hours, PaO2:FiO2<80 for 6 hours, pH<7.25 with PaCO2 >60 for >6 hours.

INTERVENTIONS:
Other: Venovenous ECMO — ECMO therapy for patients with hypoxic respiratory failure.
  Arms: Venovenous ECMO

SUMMARY:
To determine whether a strategy of adding venovenous ECMO to mechanical ventilation, as compared to mechanical ventilation alone, increases the number of intensive care free days at day 60, in patients with moderate to severe acute hypoxic respiratory failure.

DETAILED DESCRIPTION:
Mechanically ventilated patients with moderate to severe acute hypoxic respiratory failure are at increased risk of dying, short and long-term health problems and are often very costly to treat. The mechanical ventilator, whilst often lifesaving, may harm patients in two ways i) directly via damage to the lungs (termed ventilator induced lung injury), and ii) indirectly via paralysis and sedation that patients require to tolerate mechanical ventilation. Paralysis and sedation can increase the risk of secondary infections, weakness, prolonged duration of intensive care, as well as long-term physical disability. There is a need to develop new treatments that support patients and at the same time reduce these complications.

Extracorporeal membrane oxygenation (ECMO) is a device that supports the lungs by adding oxygen and removing carbon dioxide from the blood. By providing non pulmonary gas exchange, veno-venous (VV) ECMO can reduce the need for the mechanical ventilator. This in turn can reduce the risk of lung damage, and also removes the need for sedating medications so that activities like physiotherapy can begin earlier.

The REDEEM trial is a phase 2, investigator initiated, multicentre randomised controlled trial that will recruit 140 patients with moderate to severe acute hypoxic respiratory failure. It is designed to test whether adding ECMO to the mechanical ventilator, as compared to using the mechanical ventilator on its own, leads to an increase in the number of patients who survive and are discharged earlier from the intensive care unit. If the REDEEM trial confirms adding ECMO is more effective than mechanical ventilation alone, it has the potential to change the current paradigm of intensive care treatment of hypoxic respiratory failure, and could lead to changes in practice globally.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 to 65 years old
2. Acute hypoxemic respiratory failure characterised by new or worsening respiratory symptoms developing within 2 weeks prior to the onset of need for oxygen or respiratory support
3. Mechanical ventilation of <7 days
4. Moderate to severe respiratory failure, as demonstrated by two P:F ratios <150mmHg at least 6 hours apart. Arterial Blood Gases (ABG) with P:F ratio > 150mmHg are permitted between the two trial inclusion ABGs.
5. Trial of proning (unless contraindicated)

Exclusion Criteria:

1. The patient will be extubated today or tomorrow (i.e. will not remain intubated and ventilated the day after tomorrow)
2. Cardiogenic cause of respiratory failure
3. Chronic hypercapnic respiratory failure defined as PaCO2 > 60 mmHg in the outpatient setting
4. Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BIPAP used solely for sleep disordered breathing
5. Confirmed diffuse alveolar haemorrhage from vasculitis
6. Neurologic conditions, i.e. undergoing treatment for intracranial hypertension
7. Currently receiving any form of ECMO (e.g., venovenous, venoarterial, or hybrid configuration)
8. Patient needing immediate VV ECMO (as per EOLIA criteria)
9. The patient is moribund and deemed unlikely to survive past 24 hours (as determined by the clinical team)
10. The patient is being transitioned to palliative care
11. Contraindications to anticoagulation (e.g., active GI bleeding, bleeding predisposition, severe trauma)
12. Previous hypersensitivity/anaphylactic reaction to heparin or heparin-induced thrombocytopenia
13. Participation or Consent is declined, OR
14. Unable to identify or Contact surrogate decision maker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit Free days to Day 60 | 60 Days
  Days alive and free from ICU to Day 60. Day Day 0 is randomisation day, with any portion of a day is spent in an ICU counted as a day.

SECONDARY OUTCOMES:
Daily sedation scores | Day 28
  Highest (+4 Combative) and lowest (-5 Unarousable) daily Richmond Agitation and Sedation Scores (RASS). The optimal score for early mobilisation of participants on ECMO is 0 Alert and Calm.

OTHER OUTCOMES:
Extubation rates | Day 28
  Date and time of enduring extubation
Participation in early mobilisation | Day 28
  Daily assessment for mobilisation by allied health clinicians using the ICU Mobility Scale. The ICU Mobility Scale ranges from 0-Lying in Bed, to 10-Walking Independently without a Gait Aid. Score 7-Walking With the Assistance of 2 or More People is the best outcome achievable for participants on ECMO.
Number of Participants who were randomised to standard care initially and subsequently needed VV-ECMO. | Day 28
  Number of Participants who were randomised to standard care initially and subsequently needed VV-ECMO.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Day 180
  Assessment of 6 domains of functioning for participants at Day 180 follow up via telephone interview. Total possible scores are 48. A lower score indicates a better outcome.
EuroQol EQ5D-5L | Day 180
  Health-related quality of life reported via telephone interview at Day 180 using the EuroQol EQ5D. Total possible scores are 25. A lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Burrell, MBBS, Principal Investigator — Monash University
Locations (7):
- Australia (6):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Royal Prince Alfred, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
- Charite Universitatmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
The Management Committee support the view of the International Committee of Medical Journal Editors and the World Health Organisation (WHO) with reference to the ethical obligation to responsibly share data acquired by interventional clinical trials. At the conclusion of the study, the management committee will consider requests from researchers who provide a methodically sound scientific proposal as per the Data Sharing Policy set out in the Australian and New Zealand Intensive Care Research Centre (ANZIC-RC) Terms of Reference. Only de-identified data will be shared and all requests for data must comply with the ethical, regulatory, and legislative requirements governing their jurisdiction.